CLINICAL TRIAL: NCT06608316
Title: Optimizing Intermittent Theta-burst Stimulation for Enhancing Dual-Task Walking, Cognitive, and Physical Function in Mild Cognitive Impairment: a Randomized Double-Blind Controlled Trial
Brief Title: Intermittent Theta-burst Stimulation for Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Marco_PANG_2024_July
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Intermittent Theta Burst Stimulation (iTBS); Dorsolateral Prefrontal Cortex (DLPFC); dual task walking; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: After stratification according to gender and age, the participants will be randomly allocated to one of three groups: (1) Left DLPFC stimulation group, (2) Bilateral DLPFC stimulation group, and (3) Sham stimulation group, using a 1:1:1 allocation ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessors and participants were blinded to the participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Left DLPFC stimulation group (Experimental): 80% resting motor threshold (RMT) iTBS stimulated the left DLPFC 4 sessions per day at 15 min intervals (3min per session), 3 days per week for 3 weeks. Sham stimulation of the right DLPFC will be performed.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Bilateral DLPFC stimulation group (Experimental): 80% RMT iTBS stimulated the bilateral DLPFC 4 sessions per day at 15 min intervals (2 sessions on the left, 2 sessions on the right, 3 min per session), 3 days per week for 3 weeks.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Sham stimulation group (Sham Comparator): Sham coil stimulates the left and right DLPFC.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — A novel transcranial magnetic stimulation protocol called intermittent theta pulse stimulation (iTBS) effectively mimics the brain's naturally occurring theta rhythms and promotes significant synaptic changes. Compared to traditional stimulation methods, iTBS is more effective at initiating long-term potential (LTP) and produces significant excitatory effects in a shorter period of time.

SUMMARY:
The objectives of this study are to:

1. Evaluating the Impact of iTBS on Cognitive and Physical Functions: The investigators will investigate the efficacy of intermittent theta burst stimulation (iTBS) in patients with mild cognitive impairment (MCI), focusing on its effects on dual-task walking abilities, balance abilities, and cognitive function.
2. Comparing Clinical Efficacy Based on Stimulation Sites: The investigators will compare the clinical efficacy of iTBS targeting the left dorsolateral prefrontal cortex (DLPFC) versus bilateral DLPFC stimulation. This comparison aims to directly examine potential differences in therapeutic outcomes based on the site of stimulation.
3. Investigating Neurophysiological Mechanisms: The investigators plan to elucidate the neurophysiological mechanisms underlying the improvements in cognitive functions and dual-task walking abilities in MCI patients facilitated by iTBS. This will be achieved using fNIRS neuroimaging of brain activity.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) is a syndrome characterized by cognitive decline that is greater than expected with normal aging; however, it is not severe enough to meet dementia criteria. Accordingly, MCI is considered a transitional state between normal aging and dementia, with a high risk of progression to Alzheimer's disease (AD). In MCI, memory and other cognitive domains such as executive function and visuospatial skills are typically affected. Furthermore, people with MCI have impaired dual-task walking function, decreased balance, and an increased risk of falls compared to cognitively normal older adults, thus affecting the ability to perform daily activities. Moreover, sleep disturbances, such as reduced efficiency and disruptions, are common in MCI, which exacerbates cognitive decline and accelerates the progression to dementia.

Non-invasive brain stimulation (NIBS) techniques have shown potential for enhancing both cognitive and functional outcomes in neuropsychiatric diseases. Transcranial magnetic stimulation (TMS) is the most common form of NIBS, which modulates cortical excitability and neuroplasticity by inducing electromagnetic pulses in targeted brain regions. TMS can be delivered in various forms based on frequency and intervals. Intermittent theta burst stimulation (iTBS) is a type of patterned TMS that mimics endogenous theta rhythms. It has shown cognitive benefits in healthy populations as well as those with AD, depression, and other conditions, but evidence regarding its efficacy in MCI is limited.

While interventions like dual-task training and non-invasive brain stimulation (e.g., tDCS) have shown promise in mitigating dual-task coordination impairments, research specifically focusing on the impact of iTBS on dual-task walking abilities in MCI patients remains scarce. Further research is needed to explore the potential of iTBS to improve dual-task walking ability, balance, and fall prevention in MCI populations.

Although the dorsolateral prefrontal cortex (DLPFC) is often targeted with NIBS due to its role in executive functions, comparisons of bilateral versus unilateral left DLPFC stimulation have not been conducted in MCI. Overall, there is a lack of empirical evidence supporting the use of iTBS protocols to improve cognition and functional activities in MCI. Elucidating the neurophysiological mechanisms underlying NIBS techniques like iTBS remains imperative.

ELIGIBILITY:
Inclusion Criteria:

* Aged≥65 years;
* Patient-reported subjective cognitive decline and the total score of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) was between 19 and 25;
* Intact daily functioning in ADL scales and being independent in daily living, and ability to walk at least for 1 minute independently without an assistive device;
* No serious visual or hearing impairment and can complete relevant assessment and testing;
* Signed informed consent of patients and their families for iTBS treatment.

Exclusion Criteria:

* Identified with contraindications in the rTMS screening questionnaire;
* Cognitive dysfunction due to craniocerebral trauma or neurological diseases;
* Presence of severe physical illnesses such as speech disorders or unstable cardiac arrhythmias;
* Currently in a critical condition such as fever, infection, or organ failure;
* Significant damage to the left frontal lobe cortex;
* Currently taking antidepressants or psychostimulants;
* Unstable vital signs or organ failure;
* Neuropsychiatric comorbidity or affective disorder that could affect the test results;
* Patients with dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task cost in cognition (Reaction time) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Reaction time will be measured during dual-task conditions
Dual-task cost in gait (gait speed) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Gait speed under dual-task condition will be recorded
Dual-task cost in cognition (Accuracy) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Accuracy will be measured during dual-task conditions

SECONDARY OUTCOMES:
Blood oxygenation level changes of the brain | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Blood oxygenation level changes will be measured using Functional Near-Infrared Spectroscopy during dual-task conditions
Dual-task gait performance 1 (gait variability) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Gait variability will be measured during dual-task walking
Dual-task gait performance 2 (stride length) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Stride length will be measured during dual-task walking
Dual-task gait performance 3 (walking distance) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Walking distance will be measured during dual-task walking
Dual-task gait performance 4 (gait cadence) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Gait cadence will be measured during dual-task walking
Dual-task gait performance 5 (trunk stability) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Trunk stability will be measured during dual-task walking

OTHER OUTCOMES:
Hong Kong Montreal Cognitive Assessment (HK-MoCA) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Hong Kong Montreal Cognitive Assessment (HK-MoCA) will be used to global cognitive function, with total points from 0-30. Higher points indicate better performance.
N-back test | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  N-back test will be used to assess executive function.
Modified-Wisconsin Card Sorting Test | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Modified-Wisconsin Card Sorting Test will be used to assess executive function.
Hong Kong List Learning Test (HKLLT) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  The Hong Kong List Learning Test (HKLLT) will be used to assess memory function.
Brief assessment of prospective memory (short form). | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  A brief assessment of prospective memory (short form) will be used to assess memory function.
Timed Up and Go test | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Timed Up and Go test will be used used to assess mobility.
Single Leg Stance test | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Single Leg Stance test will be used used to assess balance ability.
Pittsburgh Sleep Quality Index | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. Each item is scored from 0 to 3, with a total score of 0 to 21. A higher total score indicates poorer sleep quality.
Depression, Anxiety, and Stress Scale (DASS-21) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  The Depression, Anxiety, and Stress Scale (DASS-21) will be used to assess mental health. It contains 21 items divided into three dimensions, with seven items in each dimension. Scores for each dimension range from 0 to 42, with higher scores representing higher levels of depression, anxiety, and stress.
Physical Activity Scale for the Elderly (PASE) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  The Physical Activity Scale for the Elderly (PASE) will be used to assess physical activity. There is no set range for the total PASE score; usually a higher score represents a higher level of physical activity.
Fall incidence | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Monthly telephone interviews for recording fall incidence.
Hong Kong Lawton Instrumental Activities of Daily Living Scale (HKLIADL) | before the initiation of treatment, after 3 weeks of treatment, 4 weeks after termination of the treatment
  Hong Kong Lawton Instrumental Activities of Daily Living Scale (HKLIADL) will be used to assess the ability of Instrumental Activities of Daily Living, with total points from 0-27. Higher points indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study data can be provided via contacting the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From Dec 2027 onwards
Access Criteria: By contacting the Principal Investigator (Prof. Marco PANG):
  Marco.Pang@polyu.edu.hk